CLINICAL TRIAL: NCT06198725
Title: Intervention for Children With Type 1 Diabetes Targeting Gut Microbes
Acronym: TRIM1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: Adfontes (Shanghai) Bio-technology Co.,Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Trimtab-001-01
Record Dates: First submitted 2023-12-27; First posted 2024-01-10 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes; High Fiber Diet; Beta-cell function; Gut microbiota
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High fiber intervention group (Experimental): Participants in the high fiber intervention group take high fiber dietary products (28g dietary fiber per day) for 12 weeks, and at the same time, follow the doctor's advice to use subcutaneous insulin injection for treatment.
  Interventions: Dietary Supplement: Trimtab
- Usual treatment group (No Intervention): Participants in the usual treatment group received routine diet education for diabetes and were treated with subcutaneous insulin injection according to the doctor's advice

INTERVENTIONS:
Dietary Supplement: Trimtab — High fiber group will take Trimtab (a kind of multi bran and high fiber grain compound powder) 60g per day to intake 28g dietary fiber for 12 weeks.
  Arms: High fiber intervention group

SUMMARY:
The goal of this clinical study is to evaluate the effect of nutritional intervention program based on dietary products in the clinical treatment of newly diagnosed children with type 1 diabetes. The main question aims to answer is: whether high fiber diet can protect beta-cell function in children with newly onset type 1 diabetes.

Participants will take 12 weeks of high fiber diet intervention and beta-cell function and gut microbiota structure will be analyzed.

DETAILED DESCRIPTION:
The purpose of this project is to establish an early adjuvant treatment program for children with type 1 diabetes targeting gut microbiome, and to evaluate the clinical effect and safety of a dietary product to protect the beta-cell function of newly diagnosed type 1 diabetes children and improve blood sugar control.

Plan to adopt the parallel randomized controlled clinical trial method to select newly-diagnosed type 1 diabetes children, and randomly divide them into Usual care group and High fiber diet group at a ratio of 1:1. To comprehensively evaluate the clinical effect and long-term effect of a high fiber dietary intervention product, the changes of beta-cell function, glucose metabolism, and the structure and function of gut microbiota will be compared before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as type 1 diabetes for the first time according to the diagnostic criteria of the American diabetes Association (ADA) in the past 6 months;
* One or more antibodies against GAD65, IAA, IA-2, ICA, and ZNT8 are positive;
* The daily total dose of insulin per unit weight was less than 0.5 IU/kg/day three days prior to screening;
* Fasting C-peptide (FCP)>0.1 nmol/L (0.3ng/mL);
* Age range from 6 to 12 years old;
* Have not participated in any other research projects at present;
* The guardian signs the informed consent form, the child agrees to the study, and the child over 8 years old signs the informed consent form.

Exclusion Criteria:

* Suffering from serious chronic and systemic diseases: tumors, immunodeficiency, heart failure, Cushing's syndrome, kidney diseases (including nephrotic syndrome, nephritis, glomerulonephritis, kidney stones, etc.), liver diseases (including autoimmune hepatitis, metabolic liver disease, non-alcoholic fatty liver disease, primary sclerosing cholangitis, chronic, persistent hepatitis, etc.), gallbladder diseases (including cholecystitis, gallstones, etc.), etc;
* Suffering from acute or chronic gastrointestinal diseases such as Crohn's disease, ulcerative colitis, gastroesophageal reflux disease, gastrointestinal ulcers, celiac disease, or having defecation three or more times a day in the past week or more, accompanied by watery stools;
* Blood pressure ≥ 95th percentile of the same gender, age, and height reference;
* Plasma triglycerides of 9 years and below should be ≥ 1.12mmol/L, and triglycerides of 10 years and above should be ≥ 1.46mmol/L;
* Used antibiotics within the past month for 3 days or more;
* Currently suffering from infectious diseases;
* Have the history of gastrointestinal surgery, surgery to remove appendicitis and hernia;
* Evidence of pituitary dysfunction;
* Use drugs other than insulin that can affect blood sugar levels;
* Chromosomal abnormalities (such as trisomy 21 syndrome, Turner syndrome, etc.);
* Have taken probiotics and probiotic products continuously for more than 3 days within the first month before enrollment;
* Unable to guarantee sufficient time to participate in this project.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The 2h C-peptide level of the MMTT test | 0 week and 12 weeks
  The 2-hour postprandial C-peptide is detected by the mix meal test. The C peptide level is measured using a sensitive, luminescence immunoassay, accurate to 0.01 ng/ml.

SECONDARY OUTCOMES:
Glycosylated hemoglobin level | 0 week, 4 weeks, 12 weeks and 24 weeks
  The levels of glycosylated hemoglobin is detection by high performance liquid chromatography. Accurate to 0.1%.
Glycated albumin level | 0 week, 4 weeks, 12 weeks and 24 weeks
  The levels of glycated albumin is measured by IMMULITE, accurate to 0.1%.
Fasting C peptide | 0 week, 4 weeks, 12 weeks and 24 weeks
  The level of fasting C peptide is measured using a sensitive, luminescence immunoassay, accurate to 0.01 ng/ml.
Daily insulin dosage | 0 week, 4 weeks, 12 weeks and 24 weeks
  The daily insulin dosage used per kilogram of body weight. IU/kg/d
Area under curve of blood glucose in MMTT test | 0 week and 12 weeks
  The level of blood glucose will be tested at 0 min, 30 min, 60 min and 120 min of the mix meal test, and the area under curve will be calculated.
Area under curve of C peptide in MMTT test | 0 week and 12 weeks
  The level of C peptide will be tested at 0 min, 30 min, 60 min and 120 min of the mix meal test, and the area under curve will be calculated.
Adverse event occurrence rate | 0 week, 4 weeks, 12 weeks and 24 weeks
  The incidence of all recorded adverse events
Body mass index | 0 week, 4 weeks, 12 weeks and 24 weeks
  Body mass index were calculated as weight/(height)^2.
Height | 0 week, 4 weeks, 12 weeks and 24 weeks
  Height accurate to 0.1cm
Weight | 0 week, 4 weeks, 12 weeks and 24 weeks
  Weight accurate to 0.1kg
alanine aminotransferase | 0 week, 4 weeks, 12 weeks and 24 weeks
  The level of alanine aminotransferaseis is measured by enzymatic method. Accurate to 0.01 u/l.
aspartate aminotransferase | 0 week, 4 weeks, 12 weeks and 24 weeks
  The level of aspartate aminotransferase is measured by enzymatic method. Accurate to 0.01 u/l.
Total cholesterol | 0 week, 4 weeks, 12 weeks and 24 weeks
  The level of total cholesterol is measured by enzymatic method. Accurate to 0.01 mmol/L.
Triglyceride | 0 week, 4 weeks, 12 weeks and 24 weeks
  The level of triglyceride is measured by enzymatic method. Accurate to 0.01 mmol/L.

CONTACTS AND LOCATIONS:
Overall Officials: Feihong Luo, Dr, Principal Investigator — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
The relevant data can be obtained by applying to the primary investigator